CLINICAL TRIAL: NCT03793296
Title: Percutaneous Device Closure for Significant Paravalvular Leakage After Transcatheter or Surgical Valve replacement_Pilot Study
Brief Title: Percutaneous Device Closure for Significant Paravalvular Leakage After Transcatheter or Surgical Valve Replacement
Acronym: PVL closure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: At sponsor's discretion
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2018-11
Record Dates: First submitted 2018-12-30; First posted 2019-01-04 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Valves; Heart Valve Diseases; Valvular Insufficiency
Keywords: Paravalvular leak
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paravalvular leak (Experimental): After transcatheter- or surgical valve replacement
  Interventions: Device: Percutaneous Device Closure: Vascular plug

INTERVENTIONS:
Device: Percutaneous Device Closure: Vascular plug — percutaneous transcatheter approach into cardiac valve

SUMMARY:
This study evaluates the effectiveness and safety of Percutaneous Device Closure for Significant Paravalvular Leakage after transcatheter or surgical valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Significant Paravalvular Leakage After Transcatheter or Surgical Valve Replacement
* Required treatment of paravalvular leakage due to heart failure or hemolysis
* There is a formal agreement of heart team as following

  * predicted high-risk (STS score ≥8 OR Logistic EuroSCORE ≥20% OR operative mortality is ≥15%)
* Inoperable status due to old age or frailty
* Written consent

Exclusion Criteria:

* Risk of valve embolization because of valve dehiscence or instability
* Acute myocardial ischemia (enzyme elevation, ST elevation on EKG(electrocardiogram), or chest pain/discomfort)
* Evidence of intracardiac mass, thrombus or vegetation on Transthoracic/Transesophageal echocardiographic study
* Life expectancy less than 6 months due to non-cardiac disease
* Pregnant or breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-31 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of para-valvular leakage | 1 month
  classified as none, mild, moderate or severe by doppler echocardiography according to Valve Academic Research Consortium-2(VARC-2)

SECONDARY OUTCOMES:
Event rate of all cause death | up to 5 years
Event rate of cardiac death | up to 5 years
Event rate of stroke | up to 5 years
Event rate of myocardial infarction | up to 5 years
Event rate of rehospitalization | up to 5 years
Event rate of infection | up to 5 years
  Valve related infection or infective endocarditis
Event rate of acute kidney injury | 1 month
Event rate of vascular complication | 1 month
Event rate of bleeding | 1 month
Event rate of device success | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided